CLINICAL TRIAL: NCT06227507
Title: FDA Front-of-package Pretest: High In Labels
Brief Title: High in Front-of-package Label Pretest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1641776-7
Record Dates: First submitted 2024-01-08; First posted 2024-01-29 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-01

CONDITIONS: Understanding of Food Nutrient Content

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- No icon (Experimental): Participants will be shown 3 frozen meals at once; each product will be high in 1, 2, or 3 nutrients of concern (added sugar, sodium, and/or saturated fat) and will be labeled as such with a rectangular "high in" front-of-package label. The label will solely contain "high in" and nutrient text with no icon.
  Interventions: Behavioral: Front-of-package label
- Magnifying glass (Experimental): Participants will be shown 3 frozen meals at once; each product will be high in 1, 2, or 3 nutrients of concern (added sugar, sodium, and/or saturated fat) and will be labeled as such with a rectangular "high in" front-of-package label. The label will contain "high in" and nutrient text, along with a magnifying glass icon.
  Interventions: Behavioral: Front-of-package label
- Exclamation Mark (Experimental): Participants will be shown 3 frozen meals at once; each product will be high in 1, 2, or 3 nutrients of concern (added sugar, sodium, and/or saturated fat) and will be labeled as such with a rectangular "high in" front-of-package label. The label will contain "high in" and nutrient text, along with an exclamation mark icon.
  Interventions: Behavioral: Front-of-package label
- Exclamation Mark with multiple labels (Experimental): Participants will be shown 3 frozen meals at once; each product will be high in 1, 2, or 3 nutrients of concern (added sugar, sodium, and/or saturated fat) and will be labeled as such with 1, 2, or 3 rectangular "high in" front-of-package labels, one for each specific nutrient of concern. Each label will contain "high in" and nutrient text, along with an exclamation mark icon.
  Interventions: Behavioral: Front-of-package label
- Exclamation Mark with Black Background (Experimental): Participants will be shown 3 frozen meals at once; each product will be high in 1, 2, or 3 nutrients of concern (added sugar, sodium, and/or saturated fat) and will be labeled as such with a rectangular "high in" front-of-package label. The label will contain "high in" and nutrient text, along with an exclamation mark icon. The background of the "high in" text will be black, and the "high in" text will be white.
  Interventions: Behavioral: Front-of-package label

INTERVENTIONS:
Behavioral: Front-of-package label — Participants will identify the healthfulness of three packaged foods, each displayed with front-of-package labels as specified by their assigned group.

SUMMARY:
The goal of this trial is to understand which of five "High In" front-of-package label designs is most effective at helping consumers identify the healthiest products (i.e., products that are high in the fewest number of nutrients of concern: added sugar, sodium, and saturated fat).

DETAILED DESCRIPTION:
The objective of this aim is to assess which of five "High In" front-of-package label (FOPL) designs is most effective at helping consumers identify the healthiest products (i.e., products that are high in the fewest number of nutrients of concern: added sugar, sodium, and saturated fat). The investigators will use a between-subjects randomized experiment to assess the primary outcome. Participants will be randomized to one of five label conditions modeled after the U.S. Food and Drug Administration's draft "High In" FOPL designs: 1) No Icon; 2) Magnifying Glass; 3) Exclamation Mark; 4) Exclamation Mark with multiple labels; 5) Exclamation Mark with Black Background.

The primary outcome is correct identification of the healthiest product, defined as the product that is high in the fewest nutrients of concern, including added sugars, sodium, and saturated fat (percent correct for each condition). Secondary outcomes include correct identification of which product is least healthy; which product(s) are high in added sugars, saturated fat, and sodium (3 separate questions); and perceived message effectiveness (PME) of the different labels.

Logit models will be used to compare proportions in each condition that correctly identified the items (each condition compared to every other condition). For continuous outcomes (e.g., knowledge, PME scale), the investigators will use linear regression models regressing the outcome on an indicator for experimental condition. A critical alpha 0.05 will be used, and statistical tests will be two-tailed. The Bonferroni Holm correction will be used for analyses comparing conditions 2-5 to each other for each outcome (6 comparisons).

The investigators will also measure nutrition literacy, and assess moderation on the primary outcome by nutrition literacy (continuous) and highest education attainment (Bachelor's Degree or higher vs. less than Bachelor's Degree).

ELIGIBILITY:
Inclusion Criteria:

* Equal or greater than 18 years of age
* Less than 100 years of age
* English-speaking
* U.S. residents
* Participants will reflect the U.S. Census Bureau's 2021 American Community Survey 5-year estimates for gender, race/ethnicity, educational attainment, and age

Exclusion Criteria:

* Failing the attention check question
* Completing the survey in less than 33% of the median completion time

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4052 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Identification of healthiest product - dichotomous variable "Correct" (Selected product that is high in only 1 nutrient of concern) or "Incorrect" (otherwise) | During a ~10 minute online survey
  Measured with: "Which of the products below is the healthiest in terms of added sugars, sodium, and saturated fat content? The U.S. Food and Drug Administration (FDA) recommends limiting consumption of added sugars, sodium, and saturated fat."
  There is no formal name for this measure/scale.

SECONDARY OUTCOMES:
Identification of least healthy product - dichotomous variable "Correct" (Selected product that is high in all 3 nutrients of concern) or "Incorrect" (otherwise) | During a ~10 minute online survey
  Measured with: "Which of the products below is the least healthy in terms of added sugars, sodium, and saturated fat content? The U.S. Food and Drug Administration (FDA) recommends limiting consumption of added sugars, sodium, and saturated fat."
Identification of high-sodium product(s) - dichotomous variable "Correct" (Selected all products that are high in sodium) or "Incorrect" (otherwise) | During a ~10 minute online survey
  Measured with: "Which product(s) below are high in sodium? Select all that apply."
Identification of high-saturated-fat product(s) - dichotomous variable "Correct" (Selected all products that are high in saturated fat) or "Incorrect" (otherwise) | During a ~10 minute online survey
  Measured with: "Which product(s) below are high in saturated fat? Select all that apply."
Identification of high-added-sugars product(s) - dichotomous variable "Correct" (Selected all products that are high in added sugars) or "Incorrect" (otherwise) | During a ~10 minute online survey
  Measured with: "Which product(s) below are high in added sugars? Select all that apply."
Perceived Message Effectiveness of label: Discouragement - continuous variable from a 3-item scale in which each item uses a 1-5 response scale | During a ~10 minute online survey
  Measured with discouragement item from University of North Carolina Perceived Message Effectiveness Scale: How much does this label discourage you from wanting to eat this product? Response options include Not at all, A little bit, Somewhat, Quite a bit, and A great deal.

OTHER OUTCOMES:
Nutrition literacy | During a ~10 minute online survey
  Measured with: "How confident are you that you understand Nutrition Facts labels? Below is an example of a Nutrition Facts label. [Nutrition Facts label displayed]". Response options include Not at all confident, A little confident, Somewhat confident, Very confident, and Extremely confident

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Falbe, ScD, MPH, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No